CLINICAL TRIAL: NCT02527161
Title: A Prospective, Non-randomized, Longitudinal Study of the Clinical Outcomes of Participants That Receive the Stryker Triathlon Total Knee System for Total Knee Arthroplasty Implanted Using ShapeMatch® Cutting Guides: Sub-Study B
Brief Title: Stryker Triathlon Total Knee System for Total Knee Arthroplasty Implanted Using ShapeMatch® Cutting Guides: Sub-Study B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker South Pacific (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TriShapeMatch-10_SubStudyB
Record Dates: First submitted 2015-08-03; First posted 2015-08-18 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Arthroplasties, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ShapeMatch Cutting Guides with Triathlon (Other): The ShapeMatch® Cutting Guides are intended to be used as patient-specific surgical instrumentation to assist in the positioning of knee arthroplasty components intra-operatively and in guiding the marking of bone before cutting.
  They are intended for single use only.
  Interventions: Device: ShapeMatch Cutting Guides with Triathlon

INTERVENTIONS:
Device: ShapeMatch Cutting Guides with Triathlon — All participants will undergo medical imaging assessment using Magnetic Resonance Imaging (MRI) of the affected lower limb.These images will be used to manufacture the patient-specific cutting guides for preparation of the bones prior to implantation of the total knee replacement (Pre-operatively). Patients will undergo primary total knee arthroplasty with the Triathlon® Total Knee System (Stryker Orthopaedics, Mahwah, NJ USA) using the Shapematch cutting guides to guide the bone resection. Patients will follow the standard postoperative rehabilitation program established by the investigator at each site.

SUMMARY:
This is a prospective, non-randomized, longitudinal study of the clinical outcomes of participants that receive the Stryker Triathlon® Total Knee System for Total Knee Arthroplasty implanted using ShapeMatch® Cutting Guides.

Health status and functional outcome measures will be recorded to quantify functional status of subjects before surgery and at each follow-up interval. This sub-study involved the assessment of the placement of the ShapeMatch® Cutting Guides intraoperatively and post-operatively. An assessment of post-operative patient outcomes compared to pre-operative status was also analysed.

DETAILED DESCRIPTION:
Protocol Attached in documentation.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female between the ages of 50-90.
* The patient requires a primary total knee replacement and is indicated for computer-assisted surgery.
* The patient has a primary diagnosis of osteoarthritis (OA).
* The patient has intact collateral ligaments.
* The patient is able to undergo MRI scanning of the affected limb.
* The patient has signed the study specific, HREC-approved, Informed Consent document.
* The patient is willing and able to comply with the specified pre-operative and post-operative clinical and radiographic evaluations.

Exclusion Criteria:

* The patient has a history of total, unicompartmental reconstruction or fusion of the affected joint.
* The patient has had a high tibial osteotomy or femoral osteotomy.
* The patient is morbidly obese (BMI ≥ 40).
* The patient has a deformity which will require the use of stems, wedges or augments in conjunction with the Triathlon Total Knee System.
* The patient has a varus/valgus malalignment ≥ 15° (relative to mechanical axis).
* The patient has a fixed flexion deformity ≥ 15°.
* The patient has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* The patient has a systemic or metabolic disorder leading to progressive bone deterioration.
* The patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
* The patient has a cognitive impairment, an intellectual disability or a mental illness.
* The patient is pregnant.
* The patient has metal hardware present in the region of the hip, knee or ankle (as this is known to create geometrical distortion in the region of the implant).
* The patient has any known contraindications for undergoing assessment by MRI (e.g. ferrous implants, metallic clips, magnetically activated implanted devices such as cardiac pacemakers, etc).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2018-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were assessed and then placed in either Part A or Part B. Patients in Part B were invited to participate in the extension follow-up to 5-years.
Groups:
- ShapeMatch® Cutting Guides With Triathlon®: Participants who underwent Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System using the ShapeMatch® Cutting Guides.
Period: Overall Study
Arm/Group | ShapeMatch® Cutting Guides With Triathlon®
Started | 205 (All results are reported by knee throughout record. Participant=knee.)
Completed | 73 (Completed/Not completed counts are for knees at the 5 year outcome interval.)
Not Completed | 132
Not completed — Failed MRI | 52
Not completed — Withdrawal by Subject | 19
Not completed — Delay in or unfit for surgery | 16
Not completed — MRI contraindication | 6
Not completed — Consent violation | 4
Not completed — Only Recruited to Part A | 27
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Baseline measurements are only available for participants who were invited and consented to the study.
Groups:
- ShapeMatch Cutting Guides With Triathlon: Participants who underwent Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System using the ShapeMatch® Cutting Guides.
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.04 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 62
Region of Enrollment [Number; unit: participants]
  Australia | 96

OUTCOME MEASURES:

1. Primary Outcome: Implant Location/Assessment of Alignment
Description: Implant location and limb alignment is assessed using CT scan 3 months after surgery. The mean deviation of the postoperative femoral and tibial alignment from the preoperative plan is measured in degrees.
Time Frame: 3 months Post-Operatively
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 95
degrees
  Femoral deviation pre-op to post-op | 1.70 (1.46)
  Tibial deviation pre-op to post-op | 1.91 (1.58)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)_Pain
Description: KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.)
Time Frame: Pre-operative to 5 years post-operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  Pre-op KOOS Pain score | 36.18 (17.64)
  6 weeks KOOS Pain score: number analyzed (Participants) | 99
  6 weeks KOOS Pain score | 66.23 (16.88)
  3 months KOOS Pain score | 74.96 (18.55)
  6 months KOOS Pain score: number analyzed (Participants) | 98
  6 months KOOS Pain score | 80.03 (18.12)
  1 year KOOS Pain score: number analyzed (Participants) | 76
  1 year KOOS Pain score | 85.11 (16.69)
  2 years KOOS Pain score: number analyzed (Participants) | 84
  2 years KOOS Pain score | 87.00 (18.18)
  5 years KOOS Pain score: number analyzed (Participants) | 72
  5 years KOOS Pain score | 89.58 (14.24)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks KOOS Pain; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months KOOS Pain; Test type: Superiority or Other; p = 0.0013, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KOOS Pain; Test type: Superiority; p = 0.3316, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KOOS Pain; Test type: Superiority; p = 0.3366, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year KOOS Pain; Test type: Superiority; p = 0.9826, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year KOOS Pain; Test type: Superiority; p = 0.9276, ANOVA

3. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)_Symptoms
Description: as for outcome 2
Time Frame: Pre-operative to 5 years post-operative
Population: Participants with available data. Participants=knees
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  Pre-op KOOS Symptoms | 40.94 (20.85)
  6 weeks KOOS Symptoms: number analyzed (Participants) | 99
  6 weeks KOOS Symptoms | 64.78 (16.01)
  3 months KOOS Symptoms | 71.12 (18.60)
  6 months KOOS Symptoms: number analyzed (Participants) | 99
  6 months KOOS Symptoms | 75.16 (18.54)
  1 year KOOS Symptoms: number analyzed (Participants) | 77
  1 year KOOS Symptoms | 83.12 (15.33)
  2 years KOOS Symptoms score: number analyzed (Participants) | 87
  2 years KOOS Symptoms score | 84.49 (17.07)
  5 years KOOS Symptoms: number analyzed (Participants) | 73
  5 years KOOS Symptoms | 87.90 (13.13)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks KOOS Symptoms; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months KOOS Symptoms; Test type: Superiority; p = 0.0736, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KOOS Symptoms; Test type: Superiority; p = 0.4675, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KOOS Symptoms; Test type: Superiority; p = 0.0229, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year KOOS Symptoms; Test type: Superiority; p = 0.9968, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year KOOS Symptoms; Test type: Superiority; p = 0.7761, ANOVA

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)_ADL
Description: as for outcome 2
Time Frame: Pre-operative to 5 years post-operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  Pre-op KOOS ADL: number analyzed (Participants) | 99
  Pre-op KOOS ADL | 38.08 (20.12)
  6 weeks KOOS ADL: number analyzed (Participants) | 98
  6 weeks KOOS ADL | 71.98 (17.58)
  3 months KOOS ADL | 78.75 (18.20)
  6 months KOOS ADL: number analyzed (Participants) | 99
  6 months KOOS ADL | 82.37 (17.90)
  1 year KOOS ADL: number analyzed (Participants) | 74
  1 year KOOS ADL | 88.14 (14.39)
  2 years KOOS ADL score: number analyzed (Participants) | 84
  2 years KOOS ADL score | 89.60 (15.46)
  5 years KOOS ADL score: number analyzed (Participants) | 73
  5 years KOOS ADL score | 88.80 (15.09)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks KOOS ADL; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months KOOS ADL; Test type: Superiority; p = 0.0212, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KOOS ADL; Test type: Superiority; p = 0.7173, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KOOS ADL; Test type: Superiority; p = 0.1834, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year KOOS ADL; Test type: Superiority; p = 0.9957, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KOOS ADL; Test type: Superiority; p = 0.9999, ANOVA

5. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)_S&R
Description: as for outcome 2
Time Frame: Pre-operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ShapeMatch Cutting Guides With Triathlon: The ShapeMatch® Cutting Guides are intended to be used as patient-specific surgical instrumentation to assist in the positioning of knee arthroplasty components intra-operatively and in guiding the marking of bone before cutting.
  They are intended for single use only.
  ShapeMatch Cutting Guides with Triathlon: All participants will undergo medical imaging assessment using Magnetic Resonance Imaging (MRI) of the affected lower limb.These images will be used to manufacture the patient-specific cutting guides for preparation of the bones prior to implantation of the total knee replacement (Pre-operatively). Patients will undergo primary total knee arthroplasty with the Triathlon® Total Knee System (Stryker Orthopaedics, Mahwah, NJ USA) using the Shapematch cutting guides to guide the bone resection. Patients will follow the standard postoperative rehabilitation program established by the investigator at each site.
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  Pre-op KOOS S&R: number analyzed (Participants) | 96
  Pre-op KOOS S&R | 14.45 (20.98)
  1 year KOOS S&R: number analyzed (Participants) | 65
  1 year KOOS S&R | 65.05 (25.48)
  2 years KOOS S&R: number analyzed (Participants) | 75
  2 years KOOS S&R | 65.92 (27.28)
  5 years KOOS S&R: number analyzed (Participants) | 70
  5 years KOOS S&R | 64.78 (27.00)
  6 weeks KOOS S&R: number analyzed (Participants) | 83
  6 weeks KOOS S&R | 39.06 (32.49)
  3 months KOOS S&R: number analyzed (Participants) | 89
  3 months KOOS S&R | 48.58 (28.74)
  6 months KOOS S&R: number analyzed (Participants) | 92
  6 months KOOS S&R | 58.70 (29.09)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks KOOS S&R; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months KOOS S&R; Test type: Superiority; p = 0.0522, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KOOS S&R; Test type: Superiority; p = 0.1696, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KOOS S&R; Test type: Superiority; p = 0.6942, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year KOOS S&R; Test type: Superiority; p > 0.9999, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year KOOS S&R; Test type: Superiority; p > 0.9999, ANOVA

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)_QOL
Description: as for outcome 2
Time Frame: Pre-operative to 5 years post-operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: unit of a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
unit of a scale
  Pre-op KOOS QOL | 19.92 (17.63)
  6 weeks KOOS QOL score: number analyzed (Participants) | 97
  6 weeks KOOS QOL score | 51.87 (22.12)
  3 months KOOS QOL score: number analyzed (Participants) | 99
  3 months KOOS QOL score | 61.51 (21.14)
  6 months KOOS QOL: number analyzed (Participants) | 99
  6 months KOOS QOL | 69.44 (25.39)
  1 year KOOS QOL: number analyzed (Participants) | 76
  1 year KOOS QOL | 77.09 (20.78)
  2 years KOOS QOL score: number analyzed (Participants) | 85
  2 years KOOS QOL score | 79.82 (22.53)
  5 years KOOS QOL: number analyzed (Participants) | 73
  5 years KOOS QOL | 80.19 (21.73)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks KOOS QoL; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months KOOS QoL; Test type: Superiority; p = 0.0135, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KOOS QoL; Test type: Superiority; p = 0.0829, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KOOS QoL; Test type: Superiority; p = 0.1729, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year KOOS QoL; Test type: Superiority; p = 0.9687, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year KOOS QoL; Test type: Superiority; p > 0.9999, ANOVA

7. Secondary Outcome: Short Form Health Survey 12 v2 (SF-12)_Physical Component Summary (PCS)
Description: SF-12 provides a summary measure of health status after combining the physical health score (PCS) and mental health score (MCS). The SF-12 Health Survey is a 12 item participant completed questionnaire to measure general health and well-being. It includes a physical and mental status component score: each ranging from 0 to 100 points. Low values represent a poor health state and high values represent a good health state.
Time Frame: Pre-operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  SF12 PCS Preop: number analyzed (Participants) | 95
  SF12 PCS Preop | 34.36 (7.69)
  SF12 PCS 6 weeks: number analyzed (Participants) | 95
  SF12 PCS 6 weeks | 40.27 (6.98)
  SF12 PCS 3 months: number analyzed (Participants) | 94
  SF12 PCS 3 months | 45.99 (8.09)
  SF12 PCS 6 months: number analyzed (Participants) | 93
  SF12 PCS 6 months | 47.35 (8.89)
  SF12 PCS 1 year: number analyzed (Participants) | 76
  SF12 PCS 1 year | 48.27 (8.88)
  SF12 PCS 2 years: number analyzed (Participants) | 86
  SF12 PCS 2 years | 49.90 (8.64)
  SF12 PCS 5 years: number analyzed (Participants) | 73
  SF12 PCS 5 years | 46.96 (8.66)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks SF-12 PCS; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months SF-12 PCS; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months SF-12 PCS; Test type: Superiority; p = 0.8189, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year SF-12 PCS; Test type: Superiority; p = 0.9845, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year SF-12 PCS; Test type: Superiority; p = 0.7500, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year SF-12 PCS; Test type: Superiority; p = 0.1376, ANOVA

8. Secondary Outcome: VAS Pain at Rest
Description: Pain at rest and pain during mobilization was measured using a 10 centimeter Visual analogue scale (VAS). Participants are asked to indicate their level of pain with 0 being no pain and 10 being the worst pain.
Time Frame: Pre-Operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
centimeters
  VAS pain at rest_Preop: number analyzed (Participants) | 98
  VAS pain at rest_Preop | 5.78 (2.49)
  VAS pain at rest_6 weeks: number analyzed (Participants) | 99
  VAS pain at rest_6 weeks | 3.09 (2.56)
  VAS pain at rest_3 months | 2.02 (2.14)
  VAS pain at rest_6 months: number analyzed (Participants) | 97
  VAS pain at rest_6 months | 1.45 (1.98)
  VAS pain at rest_ 1 year: number analyzed (Participants) | 77
  VAS pain at rest_ 1 year | 1.22 (1.84)
  VAS pain at rest_ 2 years: number analyzed (Participants) | 86
  VAS pain at rest_ 2 years | 1.09 (1.82)
  VAS pain at rest_ 5 years: number analyzed (Participants) | 72
  VAS pain at rest_ 5 years | 1.04 (1.65)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 week VAS Rest; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months VAS Rest; Test type: Superiority; p = 0.0031, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months VAS Rest; Test type: Superiority; p = 0.2990, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year VAS Rest; Test type: Superiority; p = 0.9832, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year VAS Rest; Test type: Superiority; p = 0.9991, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year VAS Rest; Test type: Superiority; p > 0.9999, ANOVA

9. Secondary Outcome: VAS Pain Mobilised
Description: as for outcome 8
Time Frame: Pre-Operative to 5 years post-operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units of a scale
  VAS pain during mobilization_Preop: number analyzed (Participants) | 98
  VAS pain during mobilization_Preop | 7.28 (2.07)
  VAS pain during mobilization_6 weeks: number analyzed (Participants) | 99
  VAS pain during mobilization_6 weeks | 3.47 (2.74)
  VAS pain during mobilization_3 months | 2.39 (2.48)
  VAS pain during mobilization_6 months: number analyzed (Participants) | 97
  VAS pain during mobilization_6 months | 1.83 (2.23)
  VAS pain during mobilization_1 year: number analyzed (Participants) | 77
  VAS pain during mobilization_1 year | 1.43 (1.99)
  VAS pain during mobilization_2 years: number analyzed (Participants) | 87
  VAS pain during mobilization_2 years | 1.41 (2.19)
  VAS pain during mobilization_5 years: number analyzed (Participants) | 72
  VAS pain during mobilization_5 years | 1.22 (1.92)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks VAS Mob; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months VAS Mob; Test type: Superiority; p = 0.0062, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months VAS Mob; Test type: Superiority; p = 0.3730, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year VAS Mob; Test type: Superiority; p = 0.8499, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year VAS Mob; Test type: Superiority; p > 0.9999, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year VAS Mob; Test type: Superiority; p = 0.9958, ANOVA

10. Secondary Outcome: Short Form Health Survey 12 (SF-12)_Mental Component Summary (MCS)
Description: as for outcome 7
Time Frame: Pre-operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  SF12 MCS Preop: number analyzed (Participants) | 95
  SF12 MCS Preop | 47.02 (12.49)
  SF12 MCS 6 weeks: number analyzed (Participants) | 95
  SF12 MCS 6 weeks | 49.91 (10.56)
  SF12 MCS 3 months: number analyzed (Participants) | 94
  SF12 MCS 3 months | 52.18 (9.96)
  SF12 MCS 6 months: number analyzed (Participants) | 93
  SF12 MCS 6 months | 52.58 (9.15)
  SF12 MCS 1 year: number analyzed (Participants) | 76
  SF12 MCS 1 year | 52.93 (9.28)
  SF12 MCS 2 years: number analyzed (Participants) | 86
  SF12 MCS 2 years | 52.78 (9.27)
  SF12 MCS 5 years: number analyzed (Participants) | 73
  SF12 MCS 5 years | 52.95 (10.39)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks SF-12 MCS; Test type: Superiority; p = 0.3493, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 weeks to 3 months SF-12 MCS; Test type: Superiority; p = 0.4800, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months SF-12 MCS; Test type: Superiority; p > 0.9999, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year SF-12 MCS; Test type: Superiority; p > 0.9999, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year SF-12 MCS; Test type: Superiority; p > 0.9999, ANOVA
Statistical Analysis 6: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year SF-12 MCS; Test type: Superiority; p > 0.9999, ANOVA

11. Secondary Outcome: Knee Society Clinical Rating System (KSS) Pain Scores
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a minimum score of 0 to a maximum of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: Pre-operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  KSS Pain Preop: number analyzed (Participants) | 96
  KSS Pain Preop | 32.95 (14.06)
  KSS Pain 3 months: number analyzed (Participants) | 91
  KSS Pain 3 months | 69.05 (18.46)
  KSS Pain 6 months: number analyzed (Participants) | 91
  KSS Pain 6 months | 71.36 (15.21)
  KSS Pain 1 year: number analyzed (Participants) | 83
  KSS Pain 1 year | 76.75 (16.53)
  KSS Pain 2 years: number analyzed (Participants) | 72
  KSS Pain 2 years | 78.04 (16.32)
  KSS Pain 5 years: number analyzed (Participants) | 69
  KSS Pain 5 years | 75.60 (13.96)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 6 weeks KSS Pain; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KSS Pain; Test type: Superiority; p = 0.9465, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KSS Pain; Test type: Superiority; p = 0.1215, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 years KSS Pain; Test type: Superiority; p = 0.9912, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year KSS Pain; Test type: Superiority; p = 0.8952, ANOVA

12. Secondary Outcome: Knee Society Clinical Rating System (KSS) Functional Scores
Description: as for outcome 11
Time Frame: Pre-operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  KSS functional Preop | 43.45 (19.25)
  KSS functional 3 months: number analyzed (Participants) | 99
  KSS functional 3 months | 66.82 (20.07)
  KSS functional 6 months: number analyzed (Participants) | 99
  KSS functional 6 months | 75.45 (20.28)
  KSS functional 1 year: number analyzed (Participants) | 88
  KSS functional 1 year | 76.99 (19.79)
  KSS functional 2 years: number analyzed (Participants) | 85
  KSS functional 2 years | 74.82 (23.62)
  KSS functional 5 years: number analyzed (Participants) | 71
  KSS functional 5 years | 71.44 (25.47)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 3 months KSS Function; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KSS Function; Test type: Superiority; p = 0.0266, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KSS Function; Test type: Superiority; p = 0.9880, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 years KSS Function; Test type: Superiority; p = 0.9699, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 years KSS Function; Test type: Superiority; p = 0.8575, ANOVA

13. Secondary Outcome: Knee Society Clinical Rating System (KSS) Range of Motion Scores
Description: as for outcome 11
Time Frame: Pre-operative to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  KSS ROM Preop: number analyzed (Participants) | 98
  KSS ROM Preop | 108.59 (16.74)
  KSS ROM 3 months: number analyzed (Participants) | 98
  KSS ROM 3 months | 110.40 (14.38)
  KSS ROM 6 months: number analyzed (Participants) | 96
  KSS ROM 6 months | 112.71 (12.71)
  KSS ROM 1 year: number analyzed (Participants) | 88
  KSS ROM 1 year | 115.30 (12.36)
  KSS ROM 2 years: number analyzed (Participants) | 85
  KSS ROM 2 years | 115.09 (12.40)
  KSS ROM 5 years: number analyzed (Participants) | 73
  KSS ROM 5 years | 119.11 (13.06)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from preoperative to 3 months KSS Range of Motion; Test type: Superiority; p = 0.8581, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 3 months to 6 months KSS Range of Motion; Test type: Superiority; p = 0.7664, ANOVA
Statistical Analysis 3: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 6 months to 1 year KSS Range of Motion; Test type: Superiority; p = 0.7022, ANOVA
Statistical Analysis 4: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year KSS Range of Motion; Test type: Superiority; p > 0.9999, ANOVA
Statistical Analysis 5: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year KSS Range of Motion; Test type: Superiority; p = 0.2943, ANOVA

14. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The Forgotten Joint Score is a newly-developed twelve-item, self-reported assessment of how aware recipients of hip and knee joint replacement are of their joint in everyday life. The total score for the FJS is summed, averaged then multiplied by 25 (never = 0 points; almost never = 1 point; seldom = 2 points; sometimes = 3 points; mostly = 4 points). Total score range of 0 to 100.
Time Frame: 1 to 5 years Post-Operative
Population: Participants with available data. Participants=knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ShapeMatch Cutting Guides With Triathlon
Number analyzed (Participants) | 100
units on a scale
  FJS 1 year: number analyzed (Participants) | 54
  FJS 1 year | 54.48 (30.58)
  FJS 2 years: number analyzed (Participants) | 86
  FJS 2 years | 40.28 (30.08)
  FJS 5 years: number analyzed (Participants) | 73
  FJS 5 years | 68.82 (31.17)
Statistical Analysis 1: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 1 year to 2 year Forgotten Joint Score; Test type: Superiority; p = 0.0161, ANOVA
Statistical Analysis 2: Comparison: ShapeMatch Cutting Guides With Triathlon; Change from 2 year to 5 year Forgotten Joint Score; Test type: Superiority; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | ShapeMatch Cutting Guides With Triathlon
All-Cause Mortality (participants affected / at risk) | 1/96
Serious Adverse Events (participants affected / at risk) | 48/96
Other Adverse Events (participants affected / at risk) | 47/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShapeMatch Cutting Guides With Triathlon (N=96)
Non-Operative site (Blood and lymphatic system disorders) | 2 (15)
Non-operative site (Cardiac disorders) | 5 (6)
Non-operative site (Ear and labyrinth disorders) | 2 (2)
Non-operative site (Eye disorders) | 5 (5)
Non-operative site (Gastrointestinal disorders) | 2 (2)
Non-operative site (General disorders) | 3 (3)
Non-operative site (Hepatobiliary disorders) | 1 (1)
Non-operative site (Infections and infestations) | 1 (1)
Operative site (Infections and infestations) | 2 (4)
Non-Operative site (Injury, poisoning and procedural complications) | 2 (2)
Operative Site (Injury, poisoning and procedural complications) | 4 (4)
Non-operative site (Metabolism and nutrition disorders) | 1 (1)
Non-operative site (Musculoskeletal and connective tissue disorders) | 28 (38)
Operative site (Musculoskeletal and connective tissue disorders) | 8 (8)
Non-operative site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (11)
Non-operative site (Psychiatric disorders) | 1 (1)
Non-operative site (Renal and urinary disorders) | 5 (5)
Non-operative site (Reproductive system and breast disorders) | 2 (2)
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Non-operative site (Skin and subcutaneous tissue disorders) | 3 (3)
Operative site (Skin and subcutaneous tissue disorders) | 1 (1)
Non-operative site (Surgical and medical procedures) | 22 (38)
Operative site (Surgical and medical procedures) | 6 (6)
Non-operative side (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShapeMatch Cutting Guides With Triathlon (N=96)
Non-operative site (General disorders) | 8 (10)
Non-operative site (Musculoskeletal and connective tissue disorders) | 21 (32)
Operative site (Musculoskeletal and connective tissue disorders) | 5 (9)
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Non-operative site (Skin and subcutaneous tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discloser must give at least 40 days notice to Sponsor including a copy of the proposed publication. The Sponsor can then provide comments (which Discloser is not bound to follow), request delay of publication by no more than 120 days to allow for Sponsor to protect its intellectual property, or request that the Discloser remove certain proprietary or confidential information from the study (other than the results of the study).

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-08-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02527161/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT02527161/ICF_001.pdf